CLINICAL TRIAL: NCT07298434
Title: A Phase 3, Randomized, Triple-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VYD2311 for the Prevention of COVID-19 in Adults and Adolescents
Brief Title: Study of VYD2311 for the Prevention of COVID-19
Acronym: DECLARATION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Invivyd, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VYD2311-PREV-002
Record Dates: First submitted 2025-12-18; First posted 2025-12-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: COVID-19
Keywords: COVID; COVID-19; mAb; antibody; COVID-19 prevention; VYD2311; SARS-CoV-2 Monocloncal Antibody
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VYD2311-SD (single dose) (Active Comparator): VYD2311 administered via IM injection on Day 1, followed by placebo injection (0.9% sodium chloride [normal saline]) on Day 30 and Day 60
  Interventions: Drug: VYD2311-SD
- VYD2311-MD (multidose) (Active Comparator): VYD2311 administered via IM injection on Day 1, Day 30, and Day 60
  Interventions: Drug: VYD2311-MD
- Placebo (Placebo Comparator): Normal saline administered by IM injection on Day 1, Day 30, and Day 60
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VYD2311-SD — VYD2311-SD (single-dose arm): Intramuscular injection dosing on Day 1 with VYD2311 and Intramuscular injection dosing Placebo (normal saline) on Day 30 and Day 60
  Arms: VYD2311-SD (single dose)
Drug: VYD2311-MD — VYD2311-MD (multi-dose): Intramuscular injection dosing on Day 1, Day 30, and Day 60 with VYD2311
  Arms: VYD2311-MD (multidose)
Drug: Placebo — Intramuscular injection dosing on Day 1, Day 30, and Day 60 with Placebo (Normal Saline)
  Arms: Placebo

SUMMARY:
The main purpose of this study is to test an investigational drug known as VYD2311, which is being developed to lower the risk of getting COVID-19. VYD2311 is a monoclonal antibody that attaches to the virus that causes COVID-19 and helps block it from entering your cells. It is being tested in adults and adolescents at least 12 years old. Participants in this study will be given a "study drug" that will be either VYD2311 or placebo.

The study drug will be given as a shot into the muscle in the participant's upper thigh or upper arm once a month with a total of 3 shots during the study.

This study will help researchers see how well VYD2311 works to prevent COVID-19 during the 90 days after the first shot. The study will also look at the safety and tolerability of VYD2311, how the study drug is processed by the body (pharmacokinetics), how the immune system reacts to the study drug (immunogenicity), and how well VYD2311 can block the virus from infecting cells (neutralization). To do these tests, your blood will be drawn at certain times during the study.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

1. Is an adult aged ≥18 years or an adolescent aged 12 to <18 years weighing at least 40 kg at the time of Screening. Note: Adolescent enrollment is allowed only if permitted by the local health authorities and local ethics committees.
2. Has uninterrupted access to a device (eg, mobile phone, tablet) enabled to receive study reminders (eg, SMS text messages). The parent/guardian of adolescent participants will receive the study reminders.
3. Provides written documentation of informed consent by signing a current IEC/IRB-approved ICF at the time of Screening. In the case of adolescents, parental informed consent and adolescent assent must also be obtained.
4. Is able to understand and comply with study requirements/procedures (if applicable, with assistance by a caregiver, surrogate, or LAR) based on the assessment of the Investigator.
5. For participants assigned female sex at birth:

   1. Is not of childbearing potential, OR
   2. Is of childbearing potential and practicing adequate contraception for at least 7 days before dosing on Day 1, agrees to practice adequate contraception through 6 months after any dosing, and has a negative pregnancy test result on Day 1.

Note: Pregnant participants will be eligible for enrollment after iDMC review of safety data only upon Sponsor communication to sites and only in regions permitted by local health authorities and local ethics committees. If pregnant participants are eligible for enrollment, this criterion is no longer applicable.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Prior receipt of VYD2311 or pemivibart (VYD222) within 12 months before Day 1 or plans to receive pemivibart within 90 days after Day 1.
2. Prior receipt of convalescent plasma or a mAb to SARS-CoV-2 active against currently circulating variants within 120 days before Day 1 or plans to receive convalescent plasma or an active SARS-CoV-2 mAb within 90 days after Day 1.
3. Tests positive for current SARS-CoV-2 infection by local RAT or RT-PCR on Day 1.
4. Prior known or suspected SARS-CoV-2 infection within 120 days before Day 1.
5. Exposure to someone with known or suspected SARS-CoV-2 infection in the 5 days before Day 1.
6. Is acutely ill, including symptoms suggestive of SARS-CoV-2 infection, in the opinion of the investigator or has a fever ≥38 o C (≥100.4 o F) within 3 days of Day 1.
7. Received or plans to receive a non-COVID-19 vaccine within 7 days before or after each dose of study drug.

NOTE: Other protocol defined inclusion/exclusion criteria apply

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1770 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
RT-PCR-confirmed symptomatic COVID-19 through Day 90 | 90 days

SECONDARY OUTCOMES:
Assessment of safety based on treatment-emergent adverse events, injection site reactions, and hypersensitivity reactions through Day 90 | 90 days
Serum concentrations of VYD2311 through Day 90 | 90 days
Incidence of ADAs against VYD2311 through Day 90 | 90 days
Calculated sVNA titers (VYD2311 serum concentration/variant IC50) against relevant SARS-CoV-2 variants through Day 90 | 90 days

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Invivyd Investigative Site, Long Beach, California
  - Inviviyd Investigative Site, San Diego, California
  - Invivyd Investigative Site, Orlando, Florida
  - Invivyd Investigative Site, Hinesville, Georgia
  - Invivyd Investigative Site, Melrose Park, Illinois
  - Invivyd Investigative Site, Lenexa, Kansas
  - Invivyd Investigative Site, Silver Spring, Maryland
  - Invivyd Investigative Site, Burlington, Massachusetts
  - Invivyd Investigative Site, Southfield, Michigan
  - Invivyd Investigative Site, Maplewood, Minnesota
  - Invivyd Investigative Site, Independence, Missouri
  - Invivyd Investigative Site, Jersey City, New Jersey
  - Invivyd Investigative Site, The Bronx, New York
  - Invivyd Investigative Site, Philadelphia, Pennsylvania
  - Invivyd Investigative Site, Myrtle Beach, South Carolina
  - Invivyd Investigative Site, Goodlettsville, Tennessee
  - Invivyd Investigative Site, Houston, Texas
  - Invivyd Investigative Site, Houston-2, Texas
  - Invivyd Investigative Site, Irving, Texas
  - Invivyd Investigative Site, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No